CLINICAL TRIAL: NCT04402385
Title: Aspirin to Prevent Preeclampsia in Women With Elevated Blood Pressure and Stage 1 Hypertension (ASPPIRE)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to recruit.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2000028023
Record Dates: First submitted 2020-05-22; First posted 2020-05-26 (Actual); Results first posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Pre-Eclampsia; Stage 1 Hypertension; Elevated Blood Pressure
Keywords: Aspirin
MeSH Terms: conditions — Pre-Eclampsia; Hypertension | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin (Experimental): Participants randomized to 81 mg of Aspirin daily
  Interventions: Drug: Aspirin 81 mg
- Placebo (Placebo Comparator): Participants randomized to placebo daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin 81 mg — Participants randomized to 81 mg of Aspirin daily
  Arms: Aspirin
Drug: Placebo — Participants randomized to placebo daily
  Arms: Placebo

SUMMARY:
To determine if low dose aspirin reduces the incidence of hypertensive disorders of pregnancy (gestational hypertension, preeclampsia, eclampsia, and HELLP syndrome) in pregnant women with stage 1 hypertension and elevated blood pressure.

DETAILED DESCRIPTION:
At the baseline visit, women will go through informed consent and review of study eligibility. Objectives of the study, participation requirements, eligibility inclusion and exclusion will be reviewed in detail. If these are not met, the woman is excluded from the study. If she meets inclusion criteria, a checklist of exclusion criteria will be reviewed. If any exclusions are met, the woman is excluded from the study. The consent form will be reviewed in detail. If the woman consents and signs all pages of the form, randomization follows.

Randomization will be done in a 1:1 allocation ratio between the treatment and placebo arms, stratified by blood pressure group (elevated blood pressure and stage 1 hypertension). A computer algorithm will assign participant based on random permuted blocks design with block size between 2-4 within each strata. Each participant will have an assigned Study ID number that is linked to their random assignment.

Participants will be contacted by telephone 1 week after randomization. The purpose of this visit is to ensure the participant has received study medication and initiated the regimen.

The third encounter will be 6 weeks (+/- 1week) after randomization in person to coincide with routine prenatal visit or via telephone. The purpose of this study visit is to review their pregnancy course, use of study medications, any side effects, difficulties with the study, and have opportunities to make comments and/or ask questions. The participants will be asked to bring their study medication for pill count at the time of this encounter, if the study visit is able to be performed in person. Study participants will continue their routine prenatal care with pregnancy management performed routinely per their provider.

The fourth encounter will be 16 weeks (+/- 1week) after randomization in person to coincide with routine prenatal visit or via telephone. If the participant is already delivered by this time, the visit will be performed via telephone postpartum. The purpose of this study visit is to review their pregnancy course, use of study medications, any side effects, difficulties with the study, and have opportunities to make comments and/or ask questions. The participants will be asked to bring their study medication for pill count at the time of this encounter, if the study visit is able to be performed in person.

The rest of the study will be conducted via chart review. Each prenatal visit will be reviewed for blood pressure, evaluation of symptoms, review of any laboratory and/or imaging results. New diagnoses, medications, and hospital admissions will be documented.

Delivery records will be abstracted for outcomes listed below. Neonatal records will be reviewed from birth until 1 year of age. Neonatal and infant chart abstraction will include birthweight, Apgar scores, hospital course, problem visit, diagnoses, medications, emergency department visits, and hospitalizations. Participant's postpartum course will be reviewed for 1 year postpartum, including outpatient visits, emergency department visits, and any hospitalizations.

The study will be performed by an intent-to-treat analysis. Thus, even women who discontinue study medication will be included in final analyses.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Elevated blood pressure (At least 2 systolic BP 120-129 mm Hg within 1 year pre-pregnancy until 20 weeks gestational age on at least 2 separate healthcare encounters) or Stage 1 hypertension (At least 2 systolic BP 130-139 and/or diastolic BP 80-89 within 1 year pre-pregnancy until 20 weeks gestational age on at least 2 separate healthcare encounters)
* Speaks English or Spanish
* Informed and written consent
* Confirmed single live intrauterine pregnancy (confirmed by positive cardiac motion by transvaginal or transabdominal ultrasound)

Exclusion Criteria:

* Chronic hypertension
* Pre-gestational diabetes
* Chronic renal disease

  - diagnosis of stage 1 chronic kidney disease or higher and/or GFR <60 mL/min with duration at least 3 months and/or history of kidney transplantation and/or undergoing peritoneal or hemodialysis
* Systemic lupus erythematous
* Antiphospholipid antibody syndrome (diagnosis made by having 1 or more clinical criteria and 1 or more laboratory criteria)

  * Clinical criteria: venous thrombosis, arterial thrombosis, obstetric complications (3 or more unexplained consecutive spontaneous abortions <10 weeks gestation, 1 or more unexplained deaths of a morphologically normal fetus after 10 weeks gestation, 1 or more premature births before 34 weeks gestation attributable to placental insufficiency, including severe preeclampsia or fetal growth restriction)
  * Laboratory criteria: lupus anticoagulant, anti-cardiolipin IgG or IgM with titer >99th percentile, anti-beta 2 glycoprotein IgG or IgM with titer >99th percentile. Laboratory result must be positive twice at least 12 weeks apart
* Multifetal gestation
* 20 weeks gestation at time of randomization based on American College of Obstetricians and Gynecologists dating criteria. Dating will be based on last menstrual period (LMP) if regular, sure LMP is available that agrees with ultrasound dating. Otherwise, earliest ultrasound will be used for dating purposes.
* Prior history of hypertensive disorder of pregnancy
* Current pregnancy with known chromosomal, genetic, major malformations or fetal demise, or planned termination of pregnancy
* Women with contraindications to taking aspirin (bleeding diathesis such as Von Willebrand's disease, peptic ulcer disease, aspirin hypersensitivity, nasal polyps, asthma with aspirin-induced bronchospasm, severe liver disease).
* Concurrent participation in another study that influences risk of preeclampsia
* Women who do not plan to deliver within the YNHH system

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Grechukhina, MD, Principal Investigator — Yale University; Hillart Hosier, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aspirin | Placebo
Started | 25 | 25
Completed | 20 | 19
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants from the initially enrolled that delivered successfully.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (6.4) | 29.8 (6.6) | 28.9 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 10 | 13 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 16 | 13 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Development of Hypertensive Disorder
Description: This measure is operationally defined as a yes/no response to the development of any hypertensive disorder of pregnancy (gestational hypertension, preeclampsia, eclampsia, or HELLP syndrome). This is defined by American College of Obstetricians and Gynecologists diagnostic criteria.
Time Frame: after 20 weeks gestation until 6 weeks postpartum
Population: All enrolled participants that successfully delivered.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 20 | 19
Participants
  Yes | 5 | 4
  No | 15 | 15

2. Secondary Outcome: Development of Gestational Hypertension
Description: This measure is operationally defined as a yes/no response to the development of gestational hypertension. This is defined by American College of Obstetricians and Gynecologists diagnostic criteria.
Time Frame: after 20 weeks gestation until 6 weeks postpartum
Population: All enrolled participants that successfully delivered.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 20 | 19
Participants
  Yes | 3 | 4
  No | 17 | 15

3. Secondary Outcome: Development of Preeclampsia
Description: This measure is operationally defined as a yes/no response to the development of preeclampsia. This is defined by American College of Obstetricians and Gynecologists diagnostic criteria.
Time Frame: after 20 weeks gestation until 6 weeks postpartum
Population: All enrolled participants that successfully delivered.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 20 | 19
Participants
  Yes | 2 | 0
  No | 18 | 19

4. Secondary Outcome: Development of Preeclampsia- 37 Weeks
Description: This measure is operationally defined as a yes/no response to the development of preeclampsia at less than 37 weeks of pregnancy. This is defined by American College of Obstetricians and Gynecologists diagnostic criteria.
Time Frame: up to 37 weeks gestation
Population: All enrolled participants that successfully delivered.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 20 | 19
Participants
  Yes | 0 | 0
  No | 20 | 19

5. Secondary Outcome: Development of Preeclampsia- 34 Weeks
Description: This measure is operationally defined as a yes/no response to the development of preeclampsia at less than 34 weeks of pregnancy. This is defined by American College of Obstetricians and Gynecologists diagnostic criteria.
Time Frame: up to 34 weeks gestation
Population: All enrolled participants that successfully delivered while on study.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 20 | 19
Participants
  Yes | 0 | 0
  No | 20 | 19

6. Secondary Outcome: Development of Eclampsia
Description: This measure is operationally defined as a yes/no response to the development of eclampsia. This is defined by American College of Obstetricians and Gynecologists diagnostic criteria.
Time Frame: after 20 weeks gestation until 6 weeks postpartum
Population: All enrolled participants that successfully delivered while on study.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 20 | 19
Participants
  Yes | 0 | 0
  No | 20 | 19

7. Secondary Outcome: Development of HELLP Syndrome
Description: This measure is operationally defined as a yes/no response to the development of HELLP syndrome. This is defined by American College of Obstetricians and Gynecologists diagnostic criteria.
Time Frame: after 20 weeks gestation until 6 weeks postpartum
Population: All enrolled participants that successfully delivered while on study.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 20 | 19
Participants
  Yes | 0 | 0
  No | 20 | 19

8. Secondary Outcome: Spontaneous Preterm Delivery
Description: This measure is operationally defined as a yes/no response to a spontaneous preterm delivery up to 37 weeks of pregnancy.
Time Frame: Up to 37 weeks
Population: All enrolled participants that successfully delivered while on study.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 20 | 19
Participants
  Yes | 0 | 2
  No | 20 | 17

9. Secondary Outcome: Spontaneous Preterm Delivery
Description: This measure is operationally defined as a yes/no response to a spontaneous preterm delivery up to 34 weeks of pregnancy.
Time Frame: Up to 34 weeks
Population: All enrolled participants that successfully delivered while on study.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 20 | 19
Participants
  Yes | 0 | 1
  No | 20 | 18

10. Secondary Outcome: Fetal Growth Restriction
Description: Fetal growth restriction is estimated fetal weight <10th percentile for gestational age by Hadlock criteria with Yale New Haven Health practice-specific growth curves.
Time Frame: after 20 weeks gestation until delivery
Population: All infants born to enrolled participants that successfully delivered while on study.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 20 | 19
Participants
  Yes | 0 | 2
  No | 20 | 17

11. Secondary Outcome: Birthweight
Description: Birthweight small for gestational age (<10% by sex-specific World Health Organization growth charts)
Time Frame: day of life 0
Population: All infants born from enrolled participants that successfully delivered while on study.
Measure: Mean (Standard Deviation); unit: weight in grams
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 20 | 19
weight in grams | 3320.95 (390.47) | 3271.57 (609.29)

12. Secondary Outcome: Neonatal ICU Admission
Description: Neonatal ICU admission is operationally defined as a yes/no to whether a newborn was admitted to the neonatal ICU admission.
Time Frame: Birth until 1 year of age
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 20 | 19
Participants
  NICU Admission = Yes | 1 | 3
  NICU Admission = No | 19 | 16

13. Secondary Outcome: Stillbirth
Description: Stillbirth is operationally defined as a fetal death before or during delivery (corrected when results were entered)
Time Frame: after 20 weeks gestation until delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 20 | 19
Participants
  Yes | 0 | 0
  No | 20 | 19

14. Secondary Outcome: Neonatal Adverse Events
Description: Neonatal adverse events are operationally defined as a composite yes/no response of any of the following: need for respiratory support, necrotizing enterocolitis, neonatal sepsis, retinopathy of prematurity, intraventricular hemorrhage, neonatal death.
Time Frame: Birth until 1 year of age
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 20 | 19
Participants
  Yes | 3 | 2
  No | 17 | 17

15. Secondary Outcome: Placental Abruption
Description: Placental abruption is operationally defined as a yes/no response to a placental abruption verified either clinically or as seen on pathologic placental examination.
Time Frame: after 20 weeks gestation until delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 20 | 19
Participants
  Yes | 0 | 0
  No | 20 | 19

ADVERSE EVENTS:
Time Frame: From 20 weeks gestational up to 1 year following birth
Description: Adverse event reporting only for parents that delivered while on study and their children born on study.
Groups:
- Aspirin - Parent: Participants randomized to 81 mg of Aspirin daily
  Aspirin 81 mg: Participants randomized to 81 mg of Aspirin daily
- Aspirin - Infant: Children of participants randomized to 81 mg of Aspirin daily
  Aspirin 81 mg: Participants randomized to 81 mg of Aspirin daily
- Placebo - Parent: Participants randomized to placebo daily
  Placebo: Participants randomized to placebo daily
- Placebo - Infant: Children of participants randomized to placebo daily
  Placebo: Participants randomized to placebo daily
Arm/Group | Aspirin - Parent | Aspirin - Infant | Placebo - Parent | Placebo - Infant
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/20 | 3/20 | 0/19 | 2/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin - Parent (N=20) | Aspirin - Infant (N=20) | Placebo - Parent (N=19) | Placebo - Infant (N=19)
Postpartum Hemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Microcephaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Syncytial Virus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Laryngomalacia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nosebleed (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT04402385/Prot_SAP_000.pdf